CLINICAL TRIAL: NCT04259853
Title: Quantitative Fractional Ratio-guided Non-culprit-vessel Revascularization in STEMI Patients With Multi-vessel Disease: a Prospective Multi-center Randomized Controlled Trial
Brief Title: Quantitative Fractional Ratio-guided Revascularization in STEMI Patients With Multi-vessel Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Collaborators: Pulse Medical Imaging Technology (Shanghai) Co., Ltd (Industry)
Responsible Party: Principal Investigator, Lianglong Chen, Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: the QFR-STEMI study
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: ST Elevation Myocardial Infarction; Multi-Vessel Coronary Artery Stenosis
Keywords: ST Elevation Myocardial Infarction; Multi-Vessel Coronary Artery Stenosis; Coronary physiological function; Quantitative fractional ratio; Percutaneous coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QFR-guided PCI group (Experimental): QFR-guided revascularization on non-culprit vessels in patients with STEMI
  Interventions: Procedure: PCI
- CAG-guided PCI group (Active Comparator): CAG-guided revascularization on non-culprit vessels in patients with STEMI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Revascularization on non culprit vessel

SUMMARY:
About half of patients with ST-segment elevation myocardial infarction (STEMI) have multi-vessel lesions (> 50% diameter stenosis). But how to deal with the non-culprit vessels is still controversial. Previous studies have shown that flow fractional reserve (FFR)-guided revascularization on non-culprit vessels can further improve prognosis of such patients. However, FFR requires the use of pressure guidewire and special drugs such as adenosine to maximize induction of hyperemia forcoronary artery, which will increase the cost of operation and may cause additional risks. Quantitative flow ratio (QFR) is a novel angiography-based method for deriving FFR without pressure wire or induction of hyperemia. In present, there still are poor data about QFR-guided revascularization on non-culprit vessels in patients with STEMI. The purpose of this study is to compare the clinical effects of QFR-guided with angiography-guided revascularization on non-culprit vessel in STEMI patients with multi-vessel lesions.

DETAILED DESCRIPTION:
41% -67% of patients with acute ST-segment elevation myocardial infarction (STEMI) have severe stenosis in non-culprit vessels (> 50% diameter stenosis). Compared with patients with single-vessel lesion, these patients with multi-vessel disease have a worse survival rate after percutaneous coronary intervention (PCI). Previous studies have shown that they not only receive more revascularization than the latter but also have a higher incidence of heart failure and more frequent electrical instability after myocardial infarction.

Early guidelines from European Society of Cardiology and the American College of Cardiology/American Heart Association discourage treating the non-culprit vessels in the acute phase. However, these recommendations are given mainly based on some small-sample retrospective studies.

With the use of second-generation drug-eluting stents and novel antithrombotic drugs, the clinical benefits from primary PCI and elective PCI have been greatly improved. Results from some small-sample prospective randomized studies have demonstrated that complete revascularization on STEMI patients with multi-vessel diseases is superior to a strategy of culprit-only revascularization. Especially, more recent two trials (PRAMI and CVLPRIT) further confirmed that complete revascularization in the acute phase can produce beneficial clinical results compared to culprit-only revascularization. However, stenting for these lesions in the two studies was decided based on angiographic findings regardless of whether the lesion caused myocardial ischemia or symptoms. Moreover, coronary angiography may underestimate and overestimate the functional severity of the lesion. Stent implantation preventively will lead to overtreatment, increasing additional cost and risk. Finally, not all such studies demonstrated positive findings. For example, the PRAGUE-13 study comparing angiography-guided complete revascularization with culprit-only treatment did not find that complete revascularization has more advantages. Therefore, the angiography-guided strategy for complete revascularization in STEMI patients with multi-vessel lesions remains questionable.

The clinical value of flow fractional reserve (FFR) as a gold standard for the assessment of coronary function in ischemia has been well confirmed in coronary intervention. Recently, three studies based on coronary functioning have shown that FFR-guided complete revascularization is superior to the strategy of only treating culprit lesion. However, clinical benefit of FFR is mainly from reducing the incidence of subsequent revascularization but not hard endpoints such as death. On the other hand, the time of treatment for non-culprit vessel was not completely consistent and not all patients in the FFR group received FFR measurements in these studies. Heterogeneities from these studies may weaken the clinical benefit of FFR in guiding complete revascularization in STEMI patients. Although the current guidelines recommend that non-culprit lesions be allowed for treatment when emergency PCI is performed on specific patients (Class IIa, Level A), it is still necessary to conduct studies targeted on these issues to further clarify the value of coronary functional approach in revascularization on non-culprit vessel of patients with STEMI. FFR also has certain limitations: first, FFR is an invasive test, which requires a pressure guide wire, in turn inevitably increases the cost of operation and may cause additional procedure-associated risks; secondly, drugs such as adenosine are required to maximize hyperemia of coronary artery, and these adverse drug reactions may increase the incidence of adverse clinical events, especially in the acute state of myocardial infarction.

Quantitative flow ratio (QFR) is a novel angiography-based method accurate assessing coronary physiological functions for deriving FFR without the use of pressure wire and induction of hyperemia. The three-dimensional reconstruction of the coronary arteries is performed through two angiographic images with an acquisition angle difference of > 25 °. The QFR value is finally calculated based on the flow velocity obtained by a method of frame rate counting. In the past five years, a vast number of studies confirmed QFR is highly consistent with FFR in the diagnosis of myocardial ischemia, and the diagnostic accuracy of QFR is significantly higher than that of quantitative coronary angiography. Recent studies have also shown that, compared with conventional angiography-guided PCI, QFR-guided PCI for patients with stable angina pectoris has significantly reduced adverse cardiovascular events such as death and revascularization. Especially, QFR and FFR can accurately assess the coronary physiological function status of non-culprit lesions in emergency PCI patients, and its effectiveness is consistent with FFR applied to patients with stable coronary heart disease. Although previous studies provided the theoretical support, there are still poor data on QFR-guided non-culprit revascularization on STEMI patients with multi-vessel disease. Thus, we hypothesized that strategies for QFR to assess all blood flow limiting lesions and guide revascularization during emergency PCI would lead to better short-term and long-term clinical outcomes for STEMI patients with multiple vessel lesions, including improved left ventricular function, less secondary revascularization, less frequency of hospitalization, lower medical costs.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for emergency PCI within 12 hours;
* At least one lesion with a stenosis of 50% - 90% in the non culprit vessel and PCI required by the operator.
* Voluntary acceptance of all follow-up assessments required by the protocol.
* The subject (or legal guardian) who understands the protocol requirements and treatment procedures, and signs a written informed consent before performing the examination or operation specified in the scheme.

Exclusion Criteria:

* Left main lesion (a stenosis of ≥ 50%).
* STEMI caused by stent thrombosis.
* Non culprit vessels are chronic occlusive disease (CTO).
* The anatomy of non culprit vessels not suitable for PCI.
* The TIMI flow of non culprit vessels less than grade 2.
* Patients with one of the following conditions in the treatment of infarct related vessel:

  1. Coronary artery perforation.
  2. After the treatment, there is permanent no reflow (TIMI 0-1).
  3. The stent could not be implanted.
* Patients with Killip grade III-IV who can still not tolerate PCI again after treated for one week.
* Known severe cardiac valve dysfunction requiring surgery during follow-up.
* Subjects could not tolerate dual-antiplatelet therapy.
* Woman with pregnancy or planning to pregnancy.
* Patients with known allergy to the study stent system (sirolimus, everolimus, zotarolimus) or to protocol-required concomitant medications
* Patients participating any other clinical trials.
* Expected the patients who can not be followed up regularly according to the protocol or lost during the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
NACE (Net Adverse Clinical Events) | 12 months
  A composite endpoint of all-cause mortality, recurrent myocardial infarction, any revascularization, hospitalization for heart failure, stroke, or major bleeding at 12 months.

SECONDARY OUTCOMES:
2-year NACE | 24 months
  Incidence of all-cause mortality, recurrent myocardial infarction, any revascularization, hospitalization for heart failure, stroke, or major bleeding at 24 months.
3-year NACE | 36 months
  Incidence of all-cause mortality, recurrent myocardial infarction, any revascularization, hospitalization for heart failure, stroke, or major bleeding at at 36 months.
MACE (Major Adverse Cardiovascular Events) | up to 36 months
  Incidence of composite events of cardiac death, recurrent myocardial infarction, or ischemia-driven revasculariztion at 12, 24, 36 months.

OTHER OUTCOMES:
Stent thrombosis | up to 36 months
  The incidence of stent thrombosis at 12, 24, 36 months.
Major bleeding | up to 36 months
  The incidence of bleeding at 12, 24, 36 months.
Stroke | up to 36 months
  The incidence of stroke at 12, 24, 36 months.
Cost-effective assessment | up to 12 months
  Medical costs for procedure, hospitalization, and daily medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Lianglong Chen, MD, PhD, Principal Investigator — Fujian Medical University
Locations (15):
- China (15):
  - Fuqing Hospital, Fuqing, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian provincial hospital, Fuzhou, Fujian
  - The First Hospital of Fuzhou City, Fuzhou, Fujian
  - The First Hospital of Longyan City, Longyan, Fujian
  - Ningde Hospital Affiliated to Ningde Normal University, Ningde, Fujian
  - Putian Colloge affiliated Hospital, Putian, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - QUANZHOU First Hospital, Quanzhou, Fujian
  - Sanming First Hospital, Sanming, Fujian
  - Hospital of Shaowu city, Shaowu, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Zhangzhou city's Hospital, Zhangzhou, Fujian

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corpus RA, House JA, Marso SP, Grantham JA, Huber KC Jr, Laster SB, Johnson WL, Daniels WC, Barth CW, Giorgi LV, Rutherford BD. Multivessel percutaneous coronary intervention in patients with multivessel disease and acute myocardial infarction. Am Heart J. 2004 Sep;148(3):493-500. doi: 10.1016/j.ahj.2004.03.051. PMID 15389238
- [Background] Hanratty CG, Koyama Y, Rasmussen HH, Nelson GI, Hansen PS, Ward MR. Exaggeration of nonculprit stenosis severity during acute myocardial infarction: implications for immediate multivessel revascularization. J Am Coll Cardiol. 2002 Sep 4;40(5):911-6. doi: 10.1016/s0735-1097(02)02049-1. PMID 12225715
- [Background] Janardhanan R, Kenchaiah S, Velazquez EJ, Park Y, McMurray JJ, Weaver WD, Finn PV, White HD, Marin-Neto JA, O'Connor C, Pfeffer MA, Califf RM, Solomon SD; VALIANT Investigators. Extent of coronary artery disease as a predictor of outcomes in acute myocardial infarction complicated by heart failure, left ventricular dysfunction, or both. Am Heart J. 2006 Jul;152(1):183-9. doi: 10.1016/j.ahj.2005.11.013. PMID 16824854
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Circulation. 2011 Dec 6;124(23):e574-651. doi: 10.1161/CIR.0b013e31823ba622. Epub 2011 Nov 7. No abstract available. PMID 22064601
- [Background] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578
- [Background] Stone GW, Rizvi A, Newman W, Mastali K, Wang JC, Caputo R, Doostzadeh J, Cao S, Simonton CA, Sudhir K, Lansky AJ, Cutlip DE, Kereiakes DJ; SPIRIT IV Investigators. Everolimus-eluting versus paclitaxel-eluting stents in coronary artery disease. N Engl J Med. 2010 May 6;362(18):1663-74. doi: 10.1056/NEJMoa0910496. PMID 20445180
- [Background] Montalescot G, Wiviott SD, Braunwald E, Murphy SA, Gibson CM, McCabe CH, Antman EM; TRITON-TIMI 38 investigators. Prasugrel compared with clopidogrel in patients undergoing percutaneous coronary intervention for ST-elevation myocardial infarction (TRITON-TIMI 38): double-blind, randomised controlled trial. Lancet. 2009 Feb 28;373(9665):723-31. doi: 10.1016/S0140-6736(09)60441-4. PMID 19249633
- [Background] Khattab AA, Abdel-Wahab M, Rother C, Liska B, Toelg R, Kassner G, Geist V, Richardt G. Multi-vessel stenting during primary percutaneous coronary intervention for acute myocardial infarction. A single-center experience. Clin Res Cardiol. 2008 Jan;97(1):32-8. doi: 10.1007/s00392-007-0570-4. Epub 2007 Aug 17. PMID 17694377
- [Background] Hassan A, ElGuindy A, Antoniucci D. Culprit lesion-only versus complete revascularization in patients with STEMI: Lessons learned from PRAMI, CvLPRIT, and DANAMI-3 PRIMULTI. Glob Cardiol Sci Pract. 2015 Dec 22;2015(5):60. doi: 10.5339/gcsp.2015.60. eCollection 2015. No abstract available. PMID 26925405
- [Background] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Background] Kelly DJ, McCann GP, Blackman D, Curzen NP, Dalby M, Greenwood JP, Fairbrother K, Shipley L, Kelion A, Heatherington S, Khan JN, Nazir S, Alahmar A, Flather M, Swanton H, Schofield P, Gunning M, Hall R, Gershlick AH. Complete Versus culprit-Lesion only PRimary PCI Trial (CVLPRIT): a multicentre trial testing management strategies when multivessel disease is detected at the time of primary PCI: rationale and design. EuroIntervention. 2013 Feb 22;8(10):1190-8. doi: 10.4244/EIJV8I10A183. PMID 23425543
- [Background] Hlinomaz O, Groch L, Poloková K, et al. Multivessel coronary disease diagnosed at the time of primary PCI for STEMI: complete revascularization versus conservative strategy. PRAGUE-13 trial. Kardiol Rev Int Med 2015;17:214-220.
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Background] Smits PC, Abdel-Wahab M, Neumann FJ, Boxma-de Klerk BM, Lunde K, Schotborgh CE, Piroth Z, Horak D, Wlodarczak A, Ong PJ, Hambrecht R, Angeras O, Richardt G, Omerovic E; Compare-Acute Investigators. Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction. N Engl J Med. 2017 Mar 30;376(13):1234-1244. doi: 10.1056/NEJMoa1701067. Epub 2017 Mar 18. PMID 28317428
- [Background] Mehta SR, Wood DA, Storey RF, Mehran R, Bainey KR, Nguyen H, Meeks B, Di Pasquale G, Lopez-Sendon J, Faxon DP, Mauri L, Rao SV, Feldman L, Steg PG, Avezum A, Sheth T, Pinilla-Echeverri N, Moreno R, Campo G, Wrigley B, Kedev S, Sutton A, Oliver R, Rodes-Cabau J, Stankovic G, Welsh R, Lavi S, Cantor WJ, Wang J, Nakamya J, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2019 Oct 10;381(15):1411-1421. doi: 10.1056/NEJMoa1907775. Epub 2019 Sep 1. PMID 31475795
- [Background] Kolh P, Windecker S, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A; European Society of Cardiology Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; EACTS Clinical Guidelines Committee; Sousa Uva M, Achenbach S, Pepper J, Anyanwu A, Badimon L, Bauersachs J, Baumbach A, Beygui F, Bonaros N, De Carlo M, Deaton C, Dobrev D, Dunning J, Eeckhout E, Gielen S, Hasdai D, Kirchhof P, Luckraz H, Mahrholdt H, Montalescot G, Paparella D, Rastan AJ, Sanmartin M, Sergeant P, Silber S, Tamargo J, ten Berg J, Thiele H, van Geuns RJ, Wagner HO, Wassmann S, Wendler O, Zamorano JL; Task Force on Myocardial Revascularization of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery; European Association of Percutaneous Cardiovascular Interventions. 2014 ESC/EACTS Guidelines on myocardial revascularization: the Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur J Cardiothorac Surg. 2014 Oct;46(4):517-92. doi: 10.1093/ejcts/ezu366. Epub 2014 Aug 29. No abstract available. PMID 25173601
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Background] Lauri FM, Macaya F, Mejia-Renteria H, Goto S, Yeoh J, Nakayama M, Quiros A, Liontou C, Pareek N, Fernandez-Ortiz A, Macaya C, MacCarthy P, Escaned J; Collaborators. Angiography-derived functional assessment of non-culprit coronary stenoses in primary percutaneous coronary intervention. EuroIntervention. 2020 Apr 3;15(18):e1594-e1601. doi: 10.4244/EIJ-D-18-01165. PMID 31543501